CLINICAL TRIAL: NCT01055431
Title: Teff (Eragrostis Tef) as a Functional Food for the Prevention of Pregnancy Iron-deficiency Anemia
Brief Title: A Functional Food for the Prevention of Iron-deficiency Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Manchester Metropolitan University (Other)
Responsible Party: Dr Emma Derbyshire, Manchester Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 09/H1013/69
Record Dates: First submitted 2010-01-22; First posted 2010-01-25 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Anemia
Keywords: iron; bioavailability; status; deficiency; anaemia; functional foods; child bearing
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): Control bread
  Interventions: Other: Control bread
- Teff bread (Active Comparator): Teff bread
  Interventions: Other: Teff Bread

INTERVENTIONS:
Other: Control bread — Control bread
  Other Names: Low-iron bread
  Arms: Control
Other: Teff Bread — Teff bread
  Other Names: High-iron bread
  Arms: Teff bread

SUMMARY:
It has been estimated that 1 in 2 women expecting a baby will be diagnosed with iron deficiency. In turn iron deficiency can affect the health and wellbeing or both mother and child. Studies show that low iron stores prior to conception and low iron intakes during pregnancy may both be contributing to this problem. Although dietary supplements may be one solution, research indicates that daily compliance is low (Nguyen et al., 2008). Furthermore, prescribed iron supplements may result in uncomfortable side-effects, including constipation (Wulff & Ekstrom, 2003).

It is been observed in Ethiopia that iron deficiency anemia is lower than average; a finding that has been attributed to regular "Teff" consumption (Gies et al., 2003). Teff (Eragrostis tef) is a staple food usually consumed in the form of Enjera (flat bread prepared using a range of cereals). Research has shown that Teff is a rich source of iron that is easily absorbed by the body.

Although it is believed that regular Teff consumption may prevent to onset of iron deficiency anemia there is no research to support this. Therefore, the aim of the present study is to es-tablish whether incorporating Teff into the daily diet may be one way to improve blood profile and prevent the onset of iron deficiency anemia in expectant mothers. Study findings will demonstrate whether Teff may be an alternative source of iron that can be easily incorporated into the daily diet of both pregnant mothers and the lay public.

DETAILED DESCRIPTION:
Rationale Iron deficiency anemia is considered to be one of the most prevalent forms of malnutrition in Europe (Stoltzfus, 2003 & Hercberg et al., 2001). Pregnant mothers are particularly susceptible to the onset of iron deficiency anemia (Daily & Wylie, 2008). It has been estimated that 1 in 2 pregnant women will be diagnosed with iron deficiency (Scholl, 2005). During pregnancy maternal plasma volume expands, increasing iron requirements (Scholl et al., 2000) whilst dietary intakes generally remain unchanged (Milman, 2006). Physiologically, intestinal iron absorption may increase during pregnancy but only after iron depletion has already commenced (Milman, 2006). Research strongly suggests that pregnant women are not meeting dietary guidelines for iron (Derbyshire et al., 2009).

A Sheffield (UK) study has reported that pregnant women consume around 10.2mg of iron per day (Mouratidou et al., 2006). Another investigation undertaken in a London population found that expectant mothers had a mean intake of 10.7mg iron per day (Rees et al., 2005). A further study investigating the diet of educated, Caucasian pregnant mothers reported similar figures (Derbyshire et al., 2006). Diets deficient in iron during gestation may subsequently affect infant health, in both the short and longer term (Scholl & Reilly, 2000). Iron deficiencies in pregnancy have been linked to preterm deliveries, reduced infant birth weight, length and iron stores (Daily & Wylie, 2008). Low iron stores during periods of infant brain growth may permanently impede cognitive development (Lozoff, 2007 & Lozoff & Georgieff, 2006).

Teff (Eragrostis tef) is a staple food consumed in northern, western and central Ethiopia; usually in the form of Enjera (flat bread prepared using a range of cereals, including Eragrostis tef) (Umeta et al., 2005). Research has shown that Teff is a rich source of bioavailable iron which may be attributed to its low phytate content. Bread made with Tef enjera contains around 30mg of iron per 100g and up to 35mg when the food is fermented (Umeta et al., 2005). The iron content dramatically exceeds that of common Western foods (Corn flakes 7.9mg, boiled brown rice, 0.5mg and brown bread, 2.2mg, all per 100g consumed) (FSA, 2006). Furthermore, studies have shown that the prevalence of pregnancy iron deficiency anemia is relatively low in Ethiopia (Gies et al., 2003) which may be attributed to Eragrostis tef forming a staple part of the diet (Haidar et al., 1999).

Incorporation of Teff into the daily diet of expectant mothers may help to reduce the incidence of iron-deficiency anemia. Research shows that women do not adhere to taking large tablet supplements (Nguyen et al., 2008). Teff may therefore provide an alternative source of dietary iron that can be easily incorporated into the daily diet of both pregnant mothers and the lay public.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian
* Primiparous
* Singleton pregnancy (wk 20 to wk 30)
* Non smokers
* Pre pregnancy BMI between 19.8 and 26
* Healthy, free from iron metabolism disorders (pregnancy induced hypertension
* Not taking medicines known to influence iron status
* Not taking iron supplements (multivitamins will be accounted for)
* Free from gastrointestinal disorders
* No allergies

Exclusion Criteria:

* Pregnancy haemoglobin concentrations are not within the normal range (below 70g/l or over 160g/l)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2009-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To develop Teff bread that is rich in iron (per slice). | 2 years
To establish whether iron from Teff is bioavailable. | 2 years
To conclude whether daily Teff consumption prevents iron-deficiency anemia in pregnancy. | 2 years

SECONDARY OUTCOMES:
To use a range of different biomarkers to determine iron status. | 2 years
To compare dietary intakes of iron and iron status between the Teff/control group. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr Emma J Derbyshire, Principal Investigator — Manchester Metropolitan University
Locations (1):
- Manchester Food Research Centre, Manchester Metropolitan University, Manchester, United Kingdom

REFERENCES:
- [Background] McKenna D, Spence D, Haggan SE, McCrum E, Dornan JC, Lappin TR. A randomized trial investigating an iron-rich natural mineral water as a prophylaxis against iron deficiency in pregnancy. Clin Lab Haematol. 2003 Apr;25(2):99-103. doi: 10.1046/j.1365-2257.2003.00501.x. PMID 12641613
- See also: Manchester Metropolitan University — http://mmu.ac.uk
- See also: ROCHE Foundation for Anemia Research — http://www.rofar.org